CLINICAL TRIAL: NCT03835897
Title: Breast Cancer Screening With Mammography, Ultrasound, Contrast-enhanced MRI, and Diffusion-weighted MRI in Women at High Risk for Breast Cancer
Brief Title: Breast Cancer Screening With Diffusion-weighted MRI in Women at High Risk for Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Kyung Moon, Professor, Seoul National University Hospital
Other Study IDs: Breast Screening with DWI
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective observational multicenter study to compare the outcome of breast cancer surveillance using mammography, breast US, contrast-enhanced MRI, and diffusion-weighted MR imaging (DWI) as a screening tool, in the high-risk women for breast cancer.

* Primary objective: To compare the sensitivity of mammography, breast US, contrast-enhanced MRI, and DWI for the detection of breast cancer
* Secondary objective:

  1. To compare the specificity of mammography, breast US, contrast-enhanced MRI, and DWI for the detection of breast cancer
  2. To compare the cancer detection rate of mammography, breast US, contrast-enhanced MRI, and DWI
  3. To compare the characteristics of detected cancers

DETAILED DESCRIPTION:
* Mammography, breast US, contrast-enhanced MRI, and DWI will be performed on the same day or within 1 month at baseline and then after 1 year, and images will be interpreted independently according to the Breast Imaging Reporting and Data System (BI-RADS) by experienced radiologists.
* Each eligible woman, who provides informed consent for this study, will undergo mammography, breast US, contrast-enhanced MRI, and DWI at a 3T MR scanner.
* Contrast-enhanced breast MRI will be performed before and after a gadolinium-based contrast agent injection.
* Before contrast injection, DWI with b-value of 0, 800 and 1200 s/mm2 will be performed and will transfer into the server.
* A total of 890 high-risk women for breast cancer will be enrolled in this study.
* The BI-RADS 3 or higher is defined as test-positive. The reference standard will be a biopsy or at least 1 year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 30 years and 75 years at the time of enrollment
2. Breast cancer high-risk women who meet one or more of the following criteria: 1) BRCA mutation carrier or untested first-degree relative of BRCA mutation carrier 2) Family history of breast cancer in first- or second-degree relatives and lifetime risk >20% calculated by the Tyrer-Cuzick model 3) Family history of breast cancer in first- or second-degree relatives and personal history of breast cancer 4) Lobular carcinoma in situ, atypical ductal hyperplasia, or atypical lobular hyperplasia on previous biopsy or surgery and lifetime risk >20% calculated by the Tyrer-Cuzick model 5) Thoracic radiation therapy between the ages of 10 and 30

Exclusion Criteria:

1. Women with symptoms or signs of breast cancer or recurrence
2. Women with bilateral mastectomy
3. Pregnant or lactating women
4. Women who undergo chemotherapy due to malignancy in other organs
5. In cases of contraindications to MRI using contrast media (claustrophobia, renal insufficiency GFR<30mL/min/1.73m2, metallic foreign body such as pacemaker or clips, history of severe side effects due to MR contrast agent, etc.).

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: High-risk women for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 890 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Baseline to up to 1 year
  Number of positive examinations with a tissue diagnosis of cancer within 1 year / All cancers present in the population examined in the same time period

SECONDARY OUTCOMES:
Specificity | Baseline to up to 1 year
  Number of negative examinations without tissue diagnosis of cancer within 1 year / All examinations without tissue diagnosis of cancer within the same period
Cancer detection rate (CDR) | Baseline to up to 1 year
  Number of detected cancers (invasive and in situ cancer) /1000 examinations
Biologic characteristics of breast cancer | Baseline to up to 1 year
  histologic type, tumor grade, and molecular subtype of breast cancers

CONTACTS AND LOCATIONS:
Overall Officials: Woo Kyung Moon, MD PhD, Principal Investigator — Professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shin HJ, Lee SH, Park VY, Yoon JH, Kang BJ, Yun B, Kim TH, Ko ES, Han BK, Chu AJ, Park SY, Kim HH, Moon WK. Diffusion-Weighted Magnetic Resonance Imaging for Breast Cancer Screening in High-Risk Women: Design and Imaging Protocol of a Prospective Multicenter Study in Korea. J Breast Cancer. 2021 Apr;24(2):218-228. doi: 10.4048/jbc.2021.24.e19. PMID 33913277
- [Derived] Ha SM, Chang JM, Lee SH, Kim ES, Kim SY, Kim YS, Cho N, Moon WK. Detection of Contralateral Breast Cancer Using Diffusion-Weighted Magnetic Resonance Imaging in Women with Newly Diagnosed Breast Cancer: Comparison with Combined Mammography and Whole-Breast Ultrasound. Korean J Radiol. 2021 Jun;22(6):867-879. doi: 10.3348/kjr.2020.1183. Epub 2021 Apr 1. PMID 33856137